CLINICAL TRIAL: NCT02861430
Title: Ex-vivo Sentinel Lymph Node in Stage I-II Colon Cancer: Kappa Analysis With Immunochemistry and Molecular Biology
Acronym: UNMASK
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Principal Investigator, Zaher Lakkis, MD, Centre Hospitalier Universitaire de Besancon
Other Study IDs: API-2012-30
Record Dates: First submitted 2016-08-02; First posted 2016-08-10 (Estimated); Last update posted 2025-02-11 (Actual); Status verified 2016-08

CONDITIONS: Colon Cancer; Lymph Node; Sentinel Node
Keywords: colon cancer; sentinel node
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients
  Interventions: Procedure: Immunochemistry and molecular biology on sentinel lymph node specimen

INTERVENTIONS:
Procedure: Immunochemistry and molecular biology on sentinel lymph node specimen

SUMMARY:
Unmask Trial aims to evaluate the Kappa concordance between immunochemistry and molecular biology to detecting cancer cells in sentinel lymph node in patients undergoing colectomy for non metastatic colon cancer.

ELIGIBILITY:
Inclusion Criteria:

* Colectomy for Non metastatic colon cancer

Exclusion Criteria:

* Tumor T4
* No medical insurance
* Pregnant woman
* Psychiatric disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Colon cancer
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Concordance between immunochemistry and molecular biology | 1 month
  The primary outcome is the rate of concordance between the number of positive sentinel lymph nodes detected by immunochemistry using an anti-cytokeratin antibody (KL1) and molecular biology targeting CK20 on tumoral RNA after RT-PCR.
  The rate of positivity of the sentinel lymph nodes will be then compared to the standard technique using HES coloration used in routine pathological examination.
  Only the result using the routine examination will be used to decide whether the patient should benefit from an adjuvant chemotherapy.

SECONDARY OUTCOMES:
Disease-free survival | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU Besancon, Besançon, France